CLINICAL TRIAL: NCT02921581
Title: ReIrradiation with FDG-PET Guided Dose Painting for Recurrent and Second Primary Head and Neck Cancer
Brief Title: ReIrradiation with FDG-PET Guided Dose Painting
Acronym: RIDPAINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Cancer Society (Other)
Responsible Party: Principal Investigator, Einar Dale, Senior Consultant, Oslo University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/118
Record Dates: First submitted 2016-09-27; First posted 2016-10-03 (Estimated); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Cancer
Keywords: Dose painting; 18F-FDG; Positron emission tomography; Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: FDG-PET guided dose painting

SUMMARY:
Dose-painting may increase the chance of cure at minimised radiation-induced toxicity in intensity-modulated radiotherapy (IMRT) for primary head and neck cancer. This could also apply for recurrent and second primary head and neck cancers in previously irradiated volumes. This trial (RIDPAINT) investigates the feasibility of FDG-PET guided radiotherapy using IMRT dose-painting by contours for patients with recurrent and second primary head and neck cancer.

DETAILED DESCRIPTION:
The standard re-irradiation regimen for head and neck cancer patients treated at the Oslo University Hospital is 1.5 Gy twice daily during 4 weeks with a total dose of 60 Gy.

In this study the radiotherapy is planned using 18F-FDG PET/CT making one experimental "dose-painting by contours" SIB (simultaneous integrated boost) plan with a maximum point dose of 75 Gy. The participants will be given 65 Gy and 70 Gy minimum doses to two GTVs inside the conventional GTV (60 Gy). GTV_65Gy and GTV_70Gy are determined from the SUV values from the 18F-FDG PET/CT according to the formula proposed by the Ghent group (Van der Straeten et al, R&O -06). It is expected to keep the level of normal tissue side-effects within or slightly above the level of conventional radiotherapy (i.e. maximum dose of 60 Gy). In addition to the routine follow-up, the participants will be examined with 18F-FDG PET/CT 6 months after inclusion (4 1/2 months after end of radiotherapy) and HRQL measurements.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically verified invasive carcinoma of the head and neck region; ICD10: C01, C02.0 - C02.9; C03.0 - C03.9; C04.0 - C04.9; C05.0 - C05.9; C06.0 - C06.9; C09.0 - C09.9; C10.0 - C10.9; C11.0 - C11.9; C12; C13.0 - C13.9; C14.0 - C14.9; C30; C31.0 - C31.9; C32.0 - C32.9
* Planned treatment at the Norwegian Radium Hospital or at other participating university hospitals
* Age ≥18 years
* Ability to understand and respond to the questionnaires
* Informed consent received
* Squamous cell carcinoma in the head and neck region of patients previously irradiated for head and neck cancer
* No grade 3 or more late toxicity (except xerostomia) after the initial radio(chemo)therapy
* Minimal interval 12 months after the initial radio(chemo)therapy for primary head and neck cancer
* ECOG performance status ≤ 2

Exclusion Criteria:

* Patients planned for standard curative treatment (radical RT +/-concomitant chemotherapy or postoperative RT of primary disease)
* Patients who previously have been re-irradiated for overlapping second primary or relapse
* Other second primary tumors that are not under control
* Distant metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
Number of participants accomplishing FDG-PET guided radiotherapy for recurrent and second primary head and neck cancer. | 1 month

SECONDARY OUTCOMES:
Locoregional control (at 6 months after inclusion) evaluated with PET/CT (according to RECIST). | 6 months
Number of participants with adverse events. | 3 years
  Number of participants with toxicity using CTCAE v3.0.

CONTACTS AND LOCATIONS:
Overall Officials: Einar Dale, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Skjotskift T, Evensen ME, Furre T, Moan JM, Amdal CD, Bogsrud TV, Malinen E, Dale E. Dose painting for re-irradiation of head and neck cancer. Acta Oncol. 2018 Dec;57(12):1693-1699. doi: 10.1080/0284186X.2018.1512753. Epub 2018 Oct 3. PMID 30280623